CLINICAL TRIAL: NCT05908240
Title: Prevention of Cardiovascular Disease and Mortality in Patients With Psoriasis or Psoriatic Arthritis: Translating Guidelines of Care to Better Outcomes for Patients With Psoriatic Disease
Brief Title: Prevention of Cardiovascular Disease and Mortality in Patients With Psoriasis or Psoriatic Arthritis
Acronym: CP3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Psoriasis Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 853218
Record Dates: First submitted 2023-05-25; First posted 2023-06-18 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Psoriasis; Psoriatic Arthritis; Psoriatic Conditions; Cardiovascular Diseases
MeSH Terms: conditions — Psoriasis; Arthritis, Psoriatic; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Care Coordination (Other)
  Interventions: Other: Care Coordinator Model

INTERVENTIONS:
Other: Care Coordinator Model — A centralized care coordinator at the National Psoriasis Foundation will provide evidence-based education regarding a heart healthy lifestyle (i.e., diet, exercise, smoking cessation) and guidance from the American Heart Association/American College of Cardiology regarding management of dyslipidemia and hypertension. This information will be conveyed to a primary care provider of the patient's preference.

SUMMARY:
The goal of this research is to test a novel centralized care coordinator program to assist patients with psoriatic disease in lowering their risk of cardiovascular disease through the application of standard of care approaches to improving modifiable cardiovascular risk factors.

DETAILED DESCRIPTION:
Psoriasis patients have an increased risk of cardiovascular disease and mortality but are less likely to have traditional cardiovascular risk factors identified or adequately managed. Care coordinators have previously been demonstrated to improve outcomes in patients with chronic diseases (such as comorbid diabetes and depression) and are now routinely embedded in primary care practices in integrated health systems. The goal of this research is to test a novel centralized care coordinator program to assist patients with psoriatic disease in lowering their risk of cardiovascular disease through the application of standard of care approaches to improving modifiable cardiovascular risk factors.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide informed consent
2. Male or female aged 40-75
3. Being seen by a dermatology provider in routine care for the primary encounter diagnosis of psoriasis

Exclusion Criteria:

1. Currently taking a prescription lipid lowering medication
2. Pregnant or planning pregnancy in the next 6 months
3. Has a known history of cardiovascular disease (MI, Stroke, coronary artery, cerebrovascular, or peripheral vascular disease)

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in LDL | 6 months
  Change in LDL cholesterol

SECONDARY OUTCOMES:
Addition of new medication | 6 months
  Percent newly using lipid lowering, hypertension (HTN), or diabetes (DM) medications
Change in 10-year cardiovascular (CV) risk | 6 months
  Change in predicted 10-year risk of atherosclerotic cardiovascular disease (ASCVD) among patients with baseline 10-year risk greater than or equal to 5% measured by the American College of Cardiology ASCVD risk estimator tool for predicting percent risk for atherosclerotic cardiovascular disease.
30% LDL reduction | 6 months
  Percent with 7.5% to 20% risk who achieve a 30% or greater reduction in LDL on follow up testing
50% LDL reduction | 6 months
  Percent with greater than or equal to 20% risk who achieve LDL reduction of greater than or equal to 50%
LDL reduction under 100 | 6 months
  Percent who achieve LDL less than 100 mg/dL or non-HDL less than 130 mg/dL
Change in blood pressure | 6 months
  Change in systolic blood pressure (mm Hg)
Change in cholesterol | 6 months
  Change in total cholesterol (mg/dL)
Change in HDL | 6 months
  Change in HDL cholesterol (mg/dL)
Change in non-HDL | 6 months
  Change in non-HDL cholesterol (mg/dL)
Change in HbA1c | 6 months
  Change in hemoglobin A1c level measured in percent.
Change in Weight | 6 months
  Change in weight calculated by BMI (kg/m2)
Smoking status change | 6 months
  Percent of patients who quit smoking measured by self-reported response to survey question.
Percent undergoing additional CV testing | 6 months
  Percent undergoing additional cardiovascular (CV) risk testing such as stress test, coronary calcium score or related imaging.
Change in Body Surface Area (BSA) psoriasis severity | 6 months
  Change in percent of body surface area affected by psoriasis will be assessed.
Change in Physicians Global Assessment (PGA) psoriasis severity | 6 months
  Change in PGA score measured from 0-5 with 5 being the most severe psoriasis and 0 being the least severe.
Change in dermatology life quality index (DLQI) | 6 months
  Patient reported quality of life outcomes will be assessed using DLQI. The DLQI is calculated by summing the score of 10 questions regarding impact of skin condition on daily life resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.
Change in general health | 6 months
  EQ-5D is a standardized instrument developed by the EuroQol Group as a measure of health-related quality of life that can be used in a wide range of health conditions and treatments. The EQ-5D consists of a descriptive system and the EQ VAS. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression on a scale ranging from 1 (no health state problem) to 3 (extreme health state problems). The EQ VAS records the patient's self-rated health on a vertical visual analogue scale ranging from 0, worst health state, to 100, best health state. A scoring function is used to assign a value (i.e., EQ-5D™ index score) to self-reported health states from a set of population-based preference weights. For the U.S. general population, the possible EQ-5D index scores range from -0.11 to 1.0 where 0.0 = death and 1.0 = perfect health.
Change in reported psoriasis medication use | 6 months
  Proportion of patients who have reported any change in medications taken for psoriatic disease measured through a patient reported survey.
Change in physical activity days active | 6 months
  Change in patient reported physcial activity level through the Physical Activity Questionnaire measuring the number of days active for at least 30 minutes over the past month
Change in physical activity level | 6 months
  Change in patient reported physcial activity level through the Physical Activity Questionnaire measuring the patient reported level of physical activity on a likert scale from seldom active to vigorously active.
Patient experience with Care Coordinator Model | 6 months
  Patient experience with the care coordinator will be measured through the Patient Experience Survey with a likert scale from strongly agree to strongly disagree.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Johnson Dermatology, Fort Smith, Arkansas
  - Dawes Fretzin Clinical Research, Columbus, Indiana
  - Dawes Fretzin Clinical Research, Indianapolis, Indiana
  - MiSkinCenter, Northville, Michigan
  - SUNY Downstate, Brooklyn, New York
  - City Dermatology, Bensalem, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Bellevue Dermatology Clinic, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No